CLINICAL TRIAL: NCT05954143
Title: Phase 2, Multi-Center, Randomized, Open-Label Trial of BDC-1001 as a Single Agent and in Combination With Pertuzumab in Subjects With HER2-Positive Metastatic Breast Cancer Previously Treated With Trastuzumab Deruxtecan
Brief Title: Trial of BDC-1001 +/- Pertuzumab in Subjects With HER2-Positive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Bolt Biotherapeutics, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBI-20231001
Record Dates: First submitted 2023-06-23; First posted 2023-07-20 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BDC-1001 Single Agent (Experimental): BDC-1001 administered intravenously (IV) every 2 weeks
  Interventions: Drug: BDC-1001
- BDC-1001 in Combination With Pertuzumab (Experimental): BDC-1001 administered intravenously (IV) every 2 weeks, in combination with pertuzumab administered intravenously (IV) as a fixed non-weight-based dose of 840-mg IV loading dose and then 420-mg IV maintenance dose every 3 weeks.
  Interventions: Drug: BDC-1001; Drug: Pertuzumab

INTERVENTIONS:
Drug: BDC-1001 — BDC-1001 is an immune-stimulating antibody conjugate (ISAC) designed to be delivered systemically (intravenously) and act locally by targeting HER2-expressing tumors and related metastatic disease for destruction by the innate and adaptive immune systems. BDC-1001 consists of an investigational biosimilar of the humanized monoclonal antibody (mAb) trastuzumab that is chemically conjugated to a toll-like receptor (TLR)7/8 agonist (payload) with an intervening non-cleavable, cell membrane impermeable linker.
Drug: Pertuzumab — Pertuzumab is a monoclonal antibody that targets HER2 and prevents dimerization of HER2 with other members of the HER family (HER1, HER3, and HER4), thereby blocking ligand-activated downstream signaling.
  Other Names: Perjeta®
  Arms: BDC-1001 in Combination With Pertuzumab

SUMMARY:
This is an open-label, Phase 2 study to evaluate preliminary anti-tumor activity, safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of BDC-1001 administered as a single agent and in combination with pertuzumab in subjects with human epidermal growth factor receptor 2-positive (HER2+) metastatic breast cancer (MBC) previously treated with trastuzumab deruxtecan (Enhertu®).

DETAILED DESCRIPTION:
Eligible subjects will be randomly assigned in a 1:1 ratio to receive BDC-1001 as a single agent or BDC-1001 in combination with pertuzumab. Within each treatment arm, a Simon 2-stage design will be applied. Subjects will receive study treatment (i.e., BDC-1001 or BDC-1001 in combination with pertuzumab) for up to 24 months after Cycle 1 Day 1 (C1D1), until disease progression, unacceptable toxicity, or withdrawal for any reason.

Bolt amended the protocol to transition any subjects still receiving BDC-1001 to continue receiving BDC-1001 in the Maintenance Phase. Subjects remaining on BDC-1001 will continue to receive BDC-1001 until a criterion for discontinuation has been met.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast that is HER2+ (IHC 3+ or gene amplification by ISH or NGS).
* Have received 2 or more prior lines of anti-HER2-directed therapies, at least 1 in the metastatic setting and including trastuzumab deruxtecan.
* Measurable disease as determined by RECIST v.1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Have life expectancy of greater than 12 weeks per the Investigator.
* All subjects must agree to have a biopsy prior to enrollment. If, in the judgment of the Investigator, a biopsy is not safely accessible or clinically feasible an archival tumor tissue sample must be submitted in lieu of a freshly collected specimen.

Key Exclusion Criteria:

* History of severe hypersensitivity to any ingredient of BDC-1001 or pertuzumab.
* Previous treatment with a small molecule TLR7/8 agonist or TLR7/8 agonist that has been conjugated to tumor-targeting antibody such as ISACs within 12 months before starting study treatment.
* Impaired cardiac function or history of clinically significant cardiac disease.
* Human Immunodeficiency virus (HIV) infection, active hepatitis B infection, or hepatitis C infection.
* Central nervous system metastases with the exception of disease that is asymptomatic, clinically stable, and has not required steroids for at least 28 days before starting study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bolt Clinical Development, Study Director — Bolt Biotherapeutics
Locations (4):
- United States (3):
  - City of Hope, Irvine, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Virginia Cancer Specialists, Arlington, Virginia
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled at study sites in the United States and Spain.
Groups:
- BDC-1001 Single Agent: Participants received BDC-1001 administered intravenously (IV) every 2 weeks
- BDC-1001 in Combination With Pertuzumab: Participants received BDC-1001 administered intravenously (IV) every 2 weeks, in combination with pertuzumab administered intravenously (IV) as a fixed non-weight-based dose of 840-mg IV loading dose and then 420-mg IV maintenance dose every 3 weeks.
Period: Overall Study
Arm/Group | BDC-1001 Single Agent | BDC-1001 in Combination With Pertuzumab
Started | 6 | 5
Completed | 0 | 0
Not Completed | 6 | 5
Not completed — Progressive Disease | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Study Terminated by Sponsor | 2 | 4
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BDC-1001 Single Agent | BDC-1001 in Combination With Pertuzumab | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per RECIST v1.1 as Assessed by Investigator
Description: Objective Response Rate (ORR) was defined as the proportion of participants with best overall response of confirmed Complete Response (CR) or Partial Response (PR) as determined by the treating Investigator using RECIST v1.1 criteria.
Time Frame: Up to approximately 1 year
Population: Three of the 11 participants did not have response assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | BDC-1001 Single Agent | BDC-1001 in Combination With Pertuzumab
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

2. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1 as Assessed by Investigator
Description: Duration of Response (DOR) was calculated for participants who achieved confirmed CR or PR. For such participants, DOR is defined as the duration from the start date of CR or PR (whichever response status is observed first) and subsequently confirmed, to the earliest of documented date of PD per RECIST v 1.1 or death.
  Of the 8 participants with response assessments, there were no participants with PR or CR. Because there were no responses of PR or CR, the DOR cannot be calculated.
Time Frame: Up to approximately 1 year
Population: DOR was not assessed as there were no participants with CR or PR.
Measure: Count of Participants; unit: Participants
Arm/Group | BDC-1001 Single Agent | BDC-1001 in Combination With Pertuzumab
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

3. Secondary Outcome: Disease Control Rate (DCR) Per RECIST v1.1 as Assessed by Investigator
Description: Disease Control Rate (DCR) was the proportion of participants who achieved confirmed Complete Response (CR), Partial Response (PR), or Stable Disease (SD) lasting 23 or more weeks following the first dose of study treatment.
Time Frame: Up to approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | BDC-1001 Single Agent | BDC-1001 in Combination With Pertuzumab
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

4. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST 1.1 as Assessed by Investigator
Description: Progression-free survival (PFS) was defined as the duration from the date of first study treatment administration (Cycle 1 Day 1) to the earliest date of documented PD per RECIST v1.1 or death. A death was considered a PFS event.
Time Frame: Up to approximately 1 year
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BDC-1001 Single Agent | BDC-1001 in Combination With Pertuzumab
Number analyzed (Participants) | 6 | 5
Months | 0.986 [0.427 to NA] — It was not possible to calculate the upper 95% confidence interval due to the insufficient number of participants with events. | 1.955 [1.183 to NA] — It was not possible to calculate the upper 95% confidence interval due to the insufficient number of participants with events.

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the duration from the date of first study treatment administration to the date of death, irrespective of cause.
Time Frame: Up to approximately 1 year
Population: All treated participants are included
Measure: Number; unit: Participants
Arm/Group | BDC-1001 Single Agent | BDC-1001 in Combination With Pertuzumab
Number analyzed (Participants) | 6 | 5
Participants
  Surviving at last contact before data cut off | 4 | 5
  Died due to any cause | 2 | 0

6. Secondary Outcome: Number of Participants With at Least 1 Treatment Emergent Adverse Event (TEAE)
Description: Treatment Emergent Adverse Events (TEAE) was defined as any AE that started on or after the first administration of study treatment. TEAEs were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Time Frame: Continuously from first dose of study treatment through end of treatment and Safety Follow-Up. Up to approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | BDC-1001 Single Agent | BDC-1001 in Combination With Pertuzumab
Number analyzed (Participants) | 6 | 5
Participants | 6 | 5

7. Secondary Outcome: Number of Participants Who Had Any Treatment Emergent Adverse Event (TEAE) Related to Study Treatment
Description: as for outcome 6
Time Frame: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | BDC-1001 Single Agent | BDC-1001 in Combination With Pertuzumab
Number analyzed (Participants) | 6 | 5
Participants | 3 | 5

8. Secondary Outcome: Number of Participants With Any Treatment Emergent Serious Adverse Event (SAE) Related to Study Treatment
Description: Treatment Emergent Adverse Events (TEAE) was defined as any AE that started on or after the first administration of study treatment. TEAEs were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. A Serious Adverse Event (SAE) was defined as an AE event that resulted in death, was life-threatening, required or prolongs hospitalization, caused persistent or significant disability or incapacity, resulted in congenital anomalies or birth defects, or was an important medical event.
Time Frame: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | BDC-1001 Single Agent | BDC-1001 in Combination With Pertuzumab
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up through Safety Follow-Up (up to 35 days after last dose of study treatment). This period was up to approximately 1 year.
Description: The safety population included the participants who received at least one dose of study treatment.
Arm/Group | BDC-1001 Single Agent | BDC-1001 in Combination With Pertuzumab
All-Cause Mortality (participants affected / at risk) | 2/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BDC-1001 Single Agent (N=6) | BDC-1001 in Combination With Pertuzumab (N=5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BDC-1001 Single Agent (N=6) | BDC-1001 in Combination With Pertuzumab (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 1 | 2
Fatigue (General disorders) | 3 | 3
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase (Investigations) | 0 | 1
Aspartate aminotransferase (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood lactate dehydrogenase (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Nipple exudate bloody (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Cyanosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT05954143/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT05954143/SAP_001.pdf